CLINICAL TRIAL: NCT04261127
Title: Validation of the RADIAL Algorithm for Diagnosis of Autosomal Recessive Cerebellar Ataxia
Acronym: RADIAL-VALID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7346
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Autosomal Recessive Cerebellar Ataxia
Keywords: autosomal recessive cerebellar ataxia; algorithm; genetic diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental arm (Experimental): The analysis of phenotypic data in RADIAL and the analysis of DNA (analysis of the Friedreich gene ± PMDA panel) will be performed for all patients in order to meet the main objective and the secondary objectives.
  Specifically for the secondary objectives (N ° 3, 4 and 5), randomization via eCRF (electronic case report form) will be performed for the interpretation of genetic analyzes (PMDA panel) without inducing any change for the patients. This randomization, by block and by center, will allow the attribution of one of the following two groups:
  * Control group: interpretation of genetic analyzes without the use of RADIAL;
  * Experimental group: interpretation of genetic analyzes using RADIAL.
  Genome analysis (secondary objective n ° 6) will be carried out for all the patients who remained without diagnosis at the end of the first part, and for whom the DNA of relatives is available.
  Interventions: Genetic: Genetic diagnosis (PMDA panel); Diagnostic Test: Use of RADIAL algorithm

INTERVENTIONS:
Genetic: Genetic diagnosis (PMDA panel) — Blood samples for DNA study
Diagnostic Test: Use of RADIAL algorithm — RADIAL card filling (contains clinical and biological data)

SUMMARY:
RADIAL is an algorithm which has been developed following a review of the literature on 67 autosomal recessive cerebellar ataxias (ARCA) and personal clinical experience. Frequency and specificity of each feature were defined for each autosomal recessive cerebellar ataxia, and corresponding prediction scores were assigned. Clinical and paraclinical features of patients are entered into the algorithm, and a patient's total score for each ARCA is calculated, producing a ranking of possible diagnoses. Sensitivity and specificity of the algorithm were assessed by blinded analysis of a multinational cohort of 834 patients with molecularly confirmed autosomal recessive cerebellar ataxia. The performance of the algorithm was assessed versus a blinded panel of autosomal recessive cerebellar ataxia experts. The correct diagnosis was ranked within the top 3 highest-scoring diagnoses at a sensitivity and specificity of >90% for 84% and 91% of the evaluated genes, respectively. Mean sensitivity and specificity of the top 3 highest-scoring diagnoses were 92% and 95%, respectively. Our aim is now to validate in a prospective cohort of ARCA, the performance of RADIAL to predict the correct genetic diagnosis.

ELIGIBILITY:
Inclusion Criteria:

- For patients:

1. Patient, male or female, over 5 years old (no upper age limit)
2. Patient with cerebellar ataxia who started before the age of 40
3. Patient with a family history compatible with autosomal recessive inheritance (sporadic case, consanguinity, several cases in siblings)
4. Patient in which an acquired cause of cerebellar ataxia has been excluded
5. Patient whose genetic diagnosis is unknown (NB: patients with a known negative result for the Friedreich's disease gene are eligible for inclusion))
6. For patients over 18 years old: patient speaking and reading French, able to give a signed and dated informed consent to participate in the study.

   Patients who have reached the age of majority and whose DNA has been banked and who have signed a consent form authorizing the subsequent use of this DNA for research purposes, including genetic analysis of cerebellar ataxias or associated pathologies, and for whom the RADIAL information sheet can be completed in full, are eligible for inclusion.
7. For patient under 18 years old: Tutor or person with parental authority must speak French and be able to give a signed and dated informed consent for the minor patient.

   Patients who are minors, whose DNA has been banked and for whom the parental authority has signed a consent form authorizing the subsequent use of this DNA for research purposes, including genetic analysis of cerebellar ataxias or associated pathologies, and for whom the RADIAL information sheet can be completed, are eligible.
8. Patient affiliated to the French national health insurance

   - For relatives:
9. Male or female, over 18 years old (no upper age limit)
10. Biological father or mother of a patient included in RADIAL-VALID research protocol
11. (for prospective inclusion only) To be available for a visit to the participating center where the child is being followed
12. Speaking and reading French, able to give a signed and dated informed consent to participate in the study
13. Subject affiliated to the French national health insurance

    Exclusion Criteria:

    - For patients:
14. Patient in whom targeted sequencing of a panel of PMDA genes and/or exome/genome sequencing have already been performed.

    * For patients and related:
15. Subject of a legal protection measure
16. Subject in exclusion period (determined by previous or current study)

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients for whom the final genetic diagnosis is in the top 3 of the diagnoses proposed by the RADIAL algorithm (corresponding to the diseases with the 3 highest score given by the algorithm). | At final visit (depending of genetic results from 2 to 24 month maximum after inclusion visit)
  The final diagnosis will be established after a genetic analysis and a medical interpretation of the results by geneticists.

SECONDARY OUTCOMES:
Percentage of patients for whom the final genetic diagnosis is the first diagnosis proposed by the RADIAL algorithm (corresponding to the disease with the highest score given by the algorithm). | At final visit (depending of genetic results from 2 to 24 month maximum after inclusion visit)
Comparison of interpretation times by the clinical-genetic team (genetic and clinical data) with and without the help of the RADIAL algorithm | At final visit (depending of genetic results from 2 to 24 month maximum after inclusion visit)
  Randomization is a methodological refinement that is only useful for this secondary endpoint (does not relate to the primary endpoint). The clinical and paraclinical data of all patients will be treated in the same way, and randomization concerns only the use of RADIAL made by the data biologist in sample processing. There is therefore no randomization of subjects but only of genetic results.
  At the genetic study stage (Panel PMDA panel), for the patient group randomized "with RADIAL results", the interpretation of genetic data (and in particular of the different variants found) will be done aware of the results given by RADIAL, and in the randomized group "without results RADIAL ", the analysis of the genetic data will be done in the absence of knowledge of the results provided by RADIAL.
Comparison of the satisfaction score given by the clinical-genetic team in the interpretation of data with and without the help of the RADIAL algorithm | At final visit (depending of genetic results from 2 to 24 month maximum after inclusion visit)
  Randomization is a methodological refinement that is only useful for this secondary endpoint (does not relate to the primary endpoint). The clinical and paraclinical data of all patients will be treated in the same way, and randomization concerns only the use of RADIAL made by the data biologist in sample processing. There is therefore no randomization of subjects but only of genetic results.
  At the genetic study stage (Panel PMDA panel), for the patient group randomized "with RADIAL results", the interpretation of genetic data (and in particular of the different variants found) will be done aware of the results given by RADIAL, and in the randomized group "without results RADIAL ", the analysis of the genetic data will be done in the absence of knowledge of the results provided by RADIAL.
Influence of RADIAL on genetic diagnosis: percentage of patients whose diagnosis has been reviewed after the clinical-genetic team has learned of the results proposed by RADIAL | At final visit (depending of genetic results from 2 to 24 month maximum after inclusion visit)
  Randomization is a methodological refinement that is only useful for this secondary endpoint (does not relate to the primary endpoint). The clinical and paraclinical data of all patients will be treated in the same way, and randomization concerns only the use of RADIAL made by the data biologist in sample processing. There is therefore no randomization of subjects but only of genetic results.
  At the genetic study stage (Panel PMDA panel), for the patient group randomized "with RADIAL results", the interpretation of genetic data (and in particular of the different variants found) will be done aware of the results given by RADIAL, and in the randomized group "without results RADIAL ", the analysis of the genetic data will be done in the absence of knowledge of the results provided by RADIAL.
Percentage of patients for whom the genome analysis will have detected a new gene. | At final visit (depending of genetic results from 2 to 24 month maximum after inclusion visit)
  If no diagnosis is established after the PMDA + RADIAL analyzes, additional genetic analyzes will be carried out for patient and for relatives (genome). These new analyzes should help to define the diagnosis of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Tranchant Christine, MD, Principal Investigator — CHRU Strasbourg
Locations (8):
- France (8):
  - CHU de Besancon- Neurology, Besançon
  - CHU de Dijon- Neurology, Dijon
  - CHU Lille- Neurology, Lille
  - CHU Marseille- Neurology, Marseille
  - CHU Montpellier - Neurology, Montpellier
  - CHU Nancy- Neurology, Nancy
  - CHRU de Strasbourg - Neurology/Pediatrics, Strasbourg
  - CHU Toulouse- Neurology, Toulouse

IPD SHARING:
Plan to Share IPD: No